CLINICAL TRIAL: NCT00004840
Title: Study of Antenatal Thyrotropin-Releasing Hormone in Women in Premature Labor to Prevent Lung Disease in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: Children's Hospital of Philadelphia (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 199/13784; CHP-5R01HD29201-03
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1998-10

CONDITIONS: Respiratory Distress Syndrome
Keywords: cardiovascular and respiratory diseases; neonatal disorders; rare disease; respiratory distress syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome; Respiratory Tract Diseases; Infant, Newborn, Diseases; Rare Diseases | interventions — Thyrotropin-Releasing Hormone

INTERVENTIONS:
Drug: thyrotropin-releasing hormone

SUMMARY:
OBJECTIVES:

I. Assess the efficacy and safety of antenatal administration of thyrotropin-releasing hormone to women in premature labor to improve pulmonary outcomes in preterm infants.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, double blind, multicenter study. Patients are randomized to receive antenatal thyrotropin-releasing hormone or placebo.

Patients receive thyrotropin-releasing hormone or placebo intravenously over 20 minutes every 8 hours for 4 doses.

Infants are assessed for survival and chronic lung disease until day 28 after birth, and again at 36 postmenstrual weeks.

ELIGIBILITY:
* Pregnant women in active labor with 24-29 weeks gestation
* Not eligible if any of the following is present: Bleeding Infection Hypertension (greater than 140/90 mmHg) Fetus with hydrops or life-threatening anomalies One dead fetus in multiple pregnancy

Ages: 20 Years to 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 996
Dates: Start 1998-05; Study Completion 1998-06

CONTACTS AND LOCATIONS:
Overall Officials: Roberta A. Ballard, Study Chair — Children's Hospital of Philadelphia